CLINICAL TRIAL: NCT00153049
Title: A Randomised, Double-Blind, Placebo-Controlled, 3 x 3 Factorial Trial of Telmisartan and Hydrochlorothiazide in Patients With Essential Hypertension
Brief Title: 3 x 3 Factorial Trial of Telmisartan and Hydrochlorothiazide in Patients With Essential Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 502.439
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Hydrochlorothiazide; telmisartan, hydrochlorothiazide drug combination

INTERVENTIONS:
Drug: Telmisartan
Drug: Hydrochlorothiazide
Drug: Telmisartan + Hydrochlorothiazide

SUMMARY:
1. To investigate the dose response of the combination therapy, Telmisartan and Hydrochlorothiazide for the Japanese patients with Essential Hypertension.
2. To compare this dose response with that in the US study.

DETAILED DESCRIPTION:
This is an 8-week multicentre, randomised, double-blind, double-dummy, placebo-controlled, parallel group study utilizing all cells of a 3 x 3 factorial design. Following Screening examinations and a 4-week Placebo Run-In Period, 540 patients will be randomized to receive once-daily monotherapy with either telmisartan (MICARDIS), hydrochlorothiazide, placebo, or combination therapy with telmisartan and hydrochlorothiazide for 8 weeks (Treatment Period).

This study includes nine cells, placebo, telmisartan (TEL) 40 mg, TEL 80 mg, hydrochlorothiazide (HCTZ) 6.25 mg, HCTZ 12.5 mg, TEL 40 mg/HCTZ 6.25 mg, TEL 40 mg/HCTZ 12.5 mg, TEL 80 mg/HCTZ 6.25 mg, and TEL 80 mg/HCTZ 12.5 mg.

Study Hypothesis:

The hypothesis is that the dose response model for the Japanese patient with essential hypertension which is constructed for the change of the supine diastolic blood pressure from the baseline value to end of treatment with the multiple regression analysis, is similar to that in the US study 502.204.

Comparison(s):

The primary efficacy parameter will be the change from baseline in supine diastolic blood pressure at trough (24 hours post-dose) at the last visit during the Double-Blind Period.

The dose response surface model will be constructed. The graphs of dose response surface will be generated based on the final model. The model in this study will compare with that in US study from the perspective of including the same terms in the model.

ELIGIBILITY:
Inclusion Criteria:

1. Essential hypertensive patients who meet the following criteria:

   * Mean supine DBP >= 95 and <= 114 mm Hg at each of Visits 2 and 3.
   * Mean supine DBP must not vary by more than 10 mm Hg between Visit 2 and Visit 3.
   * Mean supine systolic blood pressure (SBP) must be >= 140 and <= 200 mm Hg at Visit 3.

   (The mean DBP and SBP values are calculated as the mean of the three supine measurements taken two minutes apart.)
2. Male or female.
3. Age >= 20 and Age <= 80 years.
4. Outpatient.
5. Able to stop current antihypertensive therapy without risk to the patient.
6. Ability to provide written Informed Consent in accordance with ?Good Clinical Practice (GCP)? (MHW Ordinance No. 28, as of Mar. 27, 1997) and the local legislation.

Exclusion Criteria:

1. Known or suspected secondary hypertension (renovascular hypertension, primary aldosteronism, melanocytoma, etc.).
2. Mean supine DBP > 114 mmHg and/or mean supine SBP > 200 mmHg during any visit of the placebo run-in period.
3. Sustained ventricular tachycardia or other clinically relevant cardiac arrhythmias (atrioventricular conduction disturbance (grade II - III), atrial fibrillation etc.).
4. NYHA functional class heart failure III-IV.
5. Myocardial infarction or cardiac surgery within 6 months of signing the informed consent form.
6. Coronary artery bypass surgery or percutaneous transluminal coronary angioplasty (PTCA) within 3 months of signing the informed consent form.
7. Unstable angina within 3 months of signing the informed consent form.
8. Hypertrophic obstructive cardiomyopathy, aortic stenosis, hemodynamically relevant stenosis of aortic or mitral valve.
9. Stroke or transient ischemic attack within 6 months of signing the informed consent form.
10. History of sudden exacerbation of renal function with AT1 receptor antagonists or ACE inhibitors; post-renal transplant.
11. Patients who have previously experienced characteristic symptoms of angioedema (such as facial, tongue, pharyngeal, laryngeal swelling with dyspnea) during treatment with AT1 receptor antagonists or ACE inhibitors.
12. Known hypersensitivity to any component of the formulation, or a known hypersensitivity to sulfonamides or sulphonamide-derived drugs (e.g. thiazides).
13. Hepatic and/or renal dysfunction as defined by the following laboratory parameters:

    * SGPT(ALT) or SGOT(AST) >= 2 times the upper limit of normal at screening (Visit 1).
    * Patients who have markedly poor bile secretion by the following laboratory parameters: Patients whose direct bilirubin >= 2.0 mg/dL at screening (Visit 1).
    * Serum creatinine >= 2.1 mg/dL at screening (Visit 1).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 583 (Actual)
Dates: Start 2004-06; Primary Completion 2005-06 (Actual); Study Completion 2005-06

PRIMARY OUTCOMES:
Change from baseline in supine diastolic blood pressure (DBP) at trough (24 hours post-dose) | after 8 weeks

SECONDARY OUTCOMES:
Change in supine systolic blood pressure (SBP) at trough (24 hours post-dose) | after 8 weeks
Change in sitting systolic and diastolic blood pressure at trough (24 hours post-dose) | after 8 weeks
DBP control rate | after 8 weeks
DBP response rate | after 8 weeks
SBP response rate | after 8 weeks
Incidence of adverse events | up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Nippon Boehringer Ingelheim Co., Ltd.
Locations (21):
- Japan (21):
  - Boehringer Ingelheim Investigational Site, Annaka, Gunma
  - Boehringer Ingelheim Investigational Site, Asahi,Chiba
  - Boehringer Ingelheim Investigational Site, Fukuoka, Fukuoka
  - Boehringer Ingelheim Investigational Site, Ichinomiya, Aichi
  - Boehringer Ingelheim Investigational Site, Iida,Nagano
  - Boehringer Ingelheim Investigational Site, Inzai, Chiba
  - Boehringer Ingelheim Investigational Site, Isesaki, Gunma
  - Boehringer Ingelheim Investigational Site, Kako-gun, Hyogo
  - Boehringer Ingelheim Investigational Site, Kasuya-gun,Fukuoka
  - Boehringer Ingelheim Investigational Site, Katsushika-ku,Tokyo
  - Boehringer Ingelheim Investigational Site, Kobe, Hyogo
  - Boehringer Ingelheim Investigational Site, Koshigaya, Saitama
  - Boehringer Ingelheim Investigational Site, Mono-gun, Miyagi
  - Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - Boehringer Ingelheim Investigational Site, Sendai, Miyagi
  - Boehringer Ingelheim Investigational Site, Setagun, Gunma
  - Boehringer Ingelheim Investigational Site, Shinjyuku, Tokyo
  - Boehringer Ingelheim Investigational Site, Shiroishi, Miyagi
  - Boehringer Ingelheim Investigational Site, Suita, Osaka
  - Boehringer Ingelheim Investigational Site, Takasaki, Gunma
  - Boehringer Ingelheim Investigational Site, Taya-gun, Gunma

REFERENCES:
- [Derived] Horie Y, Higaki J, Takeuchi M. Design, statistical analysis and sample size calculation of dose response study of telmisartan and hydrochlorothiazide. Contemp Clin Trials. 2007 Sep;28(5):647-53. doi: 10.1016/j.cct.2007.02.005. Epub 2007 Feb 27. PMID 17389151